CLINICAL TRIAL: NCT00334256
Title: Phase II Trial, Multicentre, Opened Label Evaluating the Pharmacokinetics and the Safety and Toxicity of the Tenofovir-Emtricitabine Combination in Pregnant Women and Infants in Africa and Asia
Brief Title: Tenofovir/Emtricitabine for PMTCT in Africa and Asia (ANRS 12109 TEmAA)
Acronym: TEmAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12109 TEmAA
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infection; Pregnancy
Keywords: PMTCT; Resistance; HIV infection; Pregnancy
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tenofovir (TDF)
Drug: Emtricitabine (FTC)

SUMMARY:
To study the pharmacokinetic properties, safety and viral resistance pattern of the combination of tenofovir disoproxil fumarate and emtricitabine in HIV-1-infected pregnant women and their newborns, with a view to prevention of mother-to-child transmission (PMTCT) of HIV-1 in Africa and Asia.

DETAILED DESCRIPTION:
Single-dose nevirapine (sdNVP) is the option of choice for the prevention of mother-to-child transmission (PMTCT) of HIV-1 in countries with limited resources. However, the use of sdNVP results in resistance mutations with an estimated frequency at of least 15 to 70% in women at W4-W6 postpartum. These mutations could compromise the success of subsequent treatments of mother and child with antiretroviral combinations that include NVP. Pre-clinical and clinical studies suggest that a combination of TDF and FTC, drugs with interesting pharmacokinetic properties that may be a useful alternative or complement to sdNVP.

The objectives are to study the pharmacokinetic properties, safety and viral resistance pattern of the combination of tenofovir disoproxil fumarate {TDF, 600 mg} and emtricitabine {FTC, 400 mg}) in HIV-1-infected pregnant women and their newborns, with a view to prevention of mother-to-child transmission (PMTCT) of HIV-1 in Africa and Asia.

Phase II trial, multicentre, open-label will be conducted in two steps with 30 mother-infant pairs per step and with a balanced allocation in Abidjan (Côte d'Ivoire), Soweto (South Africa) and Phnom Penh (Cambodia):

Step 1: administration of TDF/FTC to the mother; Step 2: administration of TDF/FTC to the mother and the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Women received voluntary counselling and testing and knows her serological status
* HIV-1 or HIV-1+2 infection whose serological diagnosis is confirmed by two samples
* Aged 18 years or over on the day of the inclusion
* Ongoing pregnancy of between 28 and 38 weeks of gestation from the day of the inclusion. This estimate will be based on the date of the last menstruation, or ultrasound scan, or uterine height measurement
* Indication for antiretroviral treatment in the Prevention of Mother-To-Child-Transmission (PMTCT), in line with international or national recommendations in force: WHO's clinical stage 1, 2 and CD4≥200/mm3or stage 3 and CD4≥350/mm3 (No indication of antiretroviral treatment)
* Haemoglobin over 8 g/dL in the month preceding inclusion
* Blood creatinine less than three times the upper limit of normal values
* Creatinine clearance > 49 mL/min
* Transaminases (ALAT or ASAT) less than five times the upper limit of normal values
* Neutrophils ≥750/mm3
* No hypersensitivity to emtricitabine, tenofovir, tenofovir disoproxil fumarate, zidovudine, nevirapine or to the excipients
* Signed informed-consent form by the woman and, by the father of the child to be born
* Planned delivery in a hospital setting and stay for at least 72 hours afterwards
* Agreement to take no other medication during the trial without telling the investigator
* Naïve to all antiretroviral treatment and to antiretroviral prophylaxis for PMTCT during a previous pregnancy
* Permanent residence close enough to the study centre to enable follow-up as stipulated in the protocol

Exclusion Criteria:

* Under 18 years of age
* Infected by HIV-2 alone
* One of the two parents (father) refuses to sign the consent to participate (available only for Abidjan and Phnom Penh) or the mother ( for the Soweto site)
* Indication for antiretroviral treatment (stage 4 or CD4 <200/mm3 or stage 3 and CD4 <350/mm3)
* Has already taken antiretrovirals, including any exposure to previous treatment or prophylaxis for PMTCT, before inclusion in the study
* Use of drugs which can interfere with the study such as :

  * nephrotoxic drugs amphotericin B, ganciclovir, valganciclovir or cidofovir, foscarnet, aminosides, pentamidine, cisplatin
  * anticoagulants (heparin)
* Regular use of drug or alcohol
* Health problem requiring systematic treatment or hospitalization
* Severe pregnancy disease (pre-eclampsia) that is life-threatening for the mother, the infant, or for both
* Severe vomiting preventing ingestion of tablets
* Refuses to give birth at a study site and to stay in hospital for at least 72 hours afterwards
* Renal insufficiency defined by blood creatinine more than three times the upper limit of normal values
* Creatinine clearance under or equal to 49 mL/min
* Hepatic insufficiency defined by transaminases (ALAT or ASAT) more than five times the upper limit of normal values
* Neutrophils <750/mm3
* Haemoglobin <8 grams/dL in the month preceding inclusion
* Hypersensitivity to emtricitabine, tenofovir, tenofovir disoproxil fumarate, zidovudine, nevirapine or to the excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-10; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of TDF and FTC in the mother and child | during labor and first 72 hours of life

SECONDARY OUTCOMES:
Safety of TDF + FTC in pregnant women | during labor and 2 months after delivery
Safety of TDF + FTC in children | 2 months after birth
Frequency of viral resistance to TDF and FTC in the mothers and in the infected children | at D2 and W4 postpartum/postnatal
Effect of the antiretroviral combination on maternal viral load | D2 and W4 post-partum
Estimation of the mother-to-child HIV-1 transmission rate (exploratory study) | D3, W4, W6

CONTACTS AND LOCATIONS:
Overall Officials: François Dabis, MD, PhD, Study Chair — Université Bordeaux 2; Didier K Ekouevi, MD, PhD, Principal Investigator — Programme PACCI Abidjan
Locations (3):
- Calmette Hospital, Phnom Penh, Cambodia
- Centre de Prise en Charge et de Formation ACONDA, Abidjan, Côte d’Ivoire
- PHRU, Soweto, South Africa

REFERENCES:
- [Result] TEmAA ANRS 12109 Study group; Arrive E, Chaix ML, Nerrienet E, Blanche S, Rouzioux C, Coffie PA, Kruy Leang S, McIntyre J, Avit D, Srey VH, Gray G, N'Dri-Yoman T, Diallo A, Ekouevi DK, Dabis F. Tolerance and viral resistance after single-dose nevirapine with tenofovir and emtricitabine to prevent vertical transmission of HIV-1. AIDS. 2009 Apr 27;23(7):825-33. doi: 10.1097/QAD.0b013e32832949d5. PMID 19307941
- [Result] Hirt D, Urien S, Rey E, Arrive E, Ekouevi DK, Coffie P, Leang SK, Lalsab S, Avit D, Nerrienet E, McIntyre J, Blanche S, Dabis F, Treluyer JM. Population pharmacokinetics of emtricitabine in human immunodeficiency virus type 1-infected pregnant women and their neonates. Antimicrob Agents Chemother. 2009 Mar;53(3):1067-73. doi: 10.1128/AAC.00860-08. Epub 2008 Dec 22. PMID 19104016
- [Result] Hirt D, Urien S, Ekouevi DK, Rey E, Arrive E, Blanche S, Amani-Bosse C, Nerrienet E, Gray G, Kone M, Leang SK, McIntyre J, Dabis F, Treluyer JM; ANRS 12109. Population pharmacokinetics of tenofovir in HIV-1-infected pregnant women and their neonates (ANRS 12109). Clin Pharmacol Ther. 2009 Feb;85(2):182-9. doi: 10.1038/clpt.2008.201. Epub 2008 Nov 5. PMID 18987623
- See also: Sponsor web page — http://www.anrs.fr
- See also: Related Info — http://www.retroconference.org/2008/